CLINICAL TRIAL: NCT03293836
Title: Venous Ulcer: Endovenous Radiofrequency Treatment of Insufficient Perforating and Saphenous Veins Versus Multilayer Compression Bandaging - Randomized Controlled Clinical Trial
Brief Title: Venous Ulcer: Endovenous Radiofrequency Treatment Trial
Acronym: VUERT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juliana Puggina (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Juliana Puggina, MD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vuert trial; UTN (Other: U1111-1194-4910)
Record Dates: First submitted 2017-03-20; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Varicose Ulcer; Varicose Veins of Lower Limb; Saphenous Vein Injury
Keywords: Varicose ulcer; Venous ulcer; Radiofrequency ablation; Perforating veins insufficiency; Varicose veins treatment
MeSH Terms: conditions — Varicose Ulcer | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency treatment (Experimental): Radiofrequency ablation of insufficient saphenous and perforating veins plus multilayer compressive bandage treatment
  Interventions: Procedure: Radiofrequency ablation; Procedure: Multilayer Compressive Bandage
- Multilayer Compressive Bandage only (Active Comparator): Receive only compressive treatment
  Interventions: Procedure: Multilayer Compressive Bandage

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation of insufficient saphenous and perforating veins using Closure Fast and Closure Stylet catheters (medtronic)
  Arms: Radiofrequency treatment
Procedure: Multilayer Compressive Bandage — Individual receive multilayer compressive bandage once a week

SUMMARY:
The aim of this study is to analyze the effect of intravenous therapy with radiofrequency for superficial and perforating venous insufficiency versus compression therapy with multilayer banding in patients with active venous ulcer. This is a controlled, randomized prospective clinical trial. People with venous ulcers and primary venous insufficiency in superficial and perforating venous system will be studied. Participants will be divided into two experimental groups: compression therapy alone, and compression therapy associated with superficial and perforating venous system ablation. Clinical aspects, improvement in patients' quality of life and interventions cost-effectiveness will be analyzed. Patients will be followed for 12 months after ulcer healing.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years old
* venous ulcer appeared at least 4 weeks, bellow knee
* ankle-brachial index more than 0.9
* saphenous veins insufficiency plus perforating veins reflux
* saphenous vein diameter between 5 mm and 12 mm
* absence of saphenous veins thrombophlebitis
* absence of personal history of venous deep thrombosis
* absence of ultrasound evidence of actual or previous venous deep thrombosis
* absence of severe ankle anquilosis

Exclusion Criteria:

* Unable to provide informed consent
* Unable to receive surgical intervention due to severe clinical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Ulcer Healing - 12 w | 12 weeks
  Ulcers was already healed after 12 weeks
Ulcer Healing - 24 w | 24 weeks
  Ulcers was already healed after 24 weeks

SECONDARY OUTCOMES:
Ulcer Recurrence | 1 year
  Ulcer recurrence rate after 1 year of follow up
Quality of life SF-36 | at the begginning and up to 1 week after ulcer had healed
  Increasing in individual's quality of life using SF 36
Quality of life EQ- 5D | at the begginning and up to 1 week after ulcer had healed
  Increasing in individual's quality of life using EQ-5D
Quality of life VLU-Qol | at the begginning and up to 1 week after ulcer had healed
  Increasing in individual's quality of life using VLU-Qol
Quality of life CCVLUQ | at the begginning and up to 1 week after ulcer had healed
  Increasing in individual's quality of life using VLU-Qol
Health Economic Assessment | 1 year
  A cost-effectiveness analysis will be performed using the collected data of resources used in participants care along the study. Cost-utility (QALY) will be calculated using EQ-5d questionarie data

CONTACTS AND LOCATIONS:
Overall Officials: Igor R Sincos, PhD, Principal Investigator — University of Sao Paulo; Juliana Puggina, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (University of São Paulo), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puggina J, Sincos IR, Campos W Jr, Porta RMP, Dos Santos JB, De Luccia N, Puech-Leao P, Collares FB, da Silva ES. A randomized clinical trial of the effects of saphenous and perforating veins radiofrequency ablation on venous ulcer healing (VUERT trial). Phlebology. 2021 Apr;36(3):194-202. doi: 10.1177/0268355520951697. Epub 2020 Sep 14. PMID 32928070